CLINICAL TRIAL: NCT01236547
Title: A Randomized Phase II Study of Concurrent Intensity Modulated Radiation Therapy (IMRT), Paclitaxel and Pazopanib (NSC 737754)/Placebo, for the Treatment of Anaplastic Thyroid Cancer
Brief Title: Intensity-Modulated Radiation Therapy and Paclitaxel With or Without Pazopanib Hydrochloride in Treating Patients With Anaplastic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCI-2011-02614; NCI-2011-02614 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000688092; RTOG-0912 (Other: NRG Oncology); RTOG-0912 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-05

CONDITIONS: Thyroid Gland Anaplastic Carcinoma
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — Radiotherapy, Intensity-Modulated; Paclitaxel; Taxes; pazopanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (paclitaxel, pazopanib hydrochloride, IMRT) (Experimental): Patients receive paclitaxel IV over 1 hour once weekly and pazopanib hydrochloride PO QD for 2-3 weeks. Patients then receive concurrent paclitaxel IV over 1 hour once weekly and pazopanib hydrochloride PO QD for 6-7 weeks (or until radiation treatment is completed) and IMRT 5 days per week for 6.5 weeks (total of 66 Gy in 33 fractions). Beginning 25-31 days after the completion of IMRT, patients receive paclitaxel IV over 1 hour once weekly and pazopanib hydrochloride PO QD. Treatment repeats every 3 weeks for 4 cycles (for patients with no measurable disease) or continues in the absence of disease progression or unacceptable toxicity (for patients with measurable disease).
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Drug: Paclitaxel; Drug: Pazopanib Hydrochloride
- Arm II (paclitaxel, placebo, IMRT) (Active Comparator): Patients receive paclitaxel IV over 1 hour once weekly and placebo PO QD for 2-3 weeks. Patients then receive concurrent paclitaxel IV over 1 hour once weekly and placebo PO QD for 6-7 weeks (or until radiation treatment is completed) and IMRT 5 days per week for 6.5 weeks (total of 66 Gy in 33 fractions). Beginning 25-31 days after the completion of IMRT, patients receive paclitaxel IV over 1 hour once weekly and placebo PO QD. Treatment repeats every 3 weeks for 4 cycles (for patients with no measurable disease) or continues in the absence of disease progression or unacceptable toxicity (for patients with measurable disease).
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Drug: Paclitaxel; Other: Placebo Administration

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
  Arms: Arm I (paclitaxel, pazopanib hydrochloride, IMRT)
Other: Placebo Administration — Given PO
  Arms: Arm II (paclitaxel, placebo, IMRT)

SUMMARY:
This randomized phase II trial studies the side effects and how well intensity-modulated radiation therapy (IMRT) and paclitaxel with or without pazopanib hydrochloride works in treating patients with anaplastic thyroid cancer. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether radiation therapy and paclitaxel are more effective when given with pazopanib hydrochloride in treating thyroid cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of IMRT, paclitaxel, and pazopanib (pazopanib hydrochloride) suspension. (Run-in component) II. To evaluate and compare overall survival at 1 year from study registration. (Phase II component)

SECONDARY OBJECTIVES:

I. To evaluate local-regional control at 6 and 12 months. (Phase II component) II. To evaluate the rate of grade 4 (Common Terminology Criteria for Adverse Events version 4.0 [CTCAE, v. 4.0]) hemorrhage, grade 4 febrile neutropenia, or any grade 5 adverse event assessed to be definitely, probably, or possibly related to the induction or concurrent treatment components of the protocol regimen. (Phase II component) III. To evaluate the rates of other adverse events (CTCAE, v. 4.0) assessed to be definitely, probably, or possibly related to the induction or concurrent treatment components of the protocol regimen. (Phase II component) IV. To evaluate the rate of treatment discontinuation due to toxicity during the induction or concurrent treatment components of the protocol regimen. (Phase II component) V. To evaluate response (as per Response Evaluation Criteria in Solid Tumors [RECIST]) of the primary site following the treatment component in subjects with measurable disease prior to chemoradiation. (Phase II component)

OUTLINE:

RUN-IN COMPONENT: Patients receive paclitaxel intravenously (IV) over 1 hour once weekly and pazopanib hydrochloride orally (PO) once daily (QD) for 2-3 weeks. Patients then receive concurrent paclitaxel IV over 1 hour once weekly and pazopanib hydrochloride PO QD for 6-7 weeks (or until radiation treatment is completed) and intensity-modulated radiotherapy (IMRT) 5 days per week for 6.5 weeks (total of 66 Gy in 33 fractions). Beginning 25-31 days after the completion of IMRT, patients receive paclitaxel IV over 1 hour once weekly and pazopanib hydrochloride PO QD. Treatment repeats every 3 weeks for 4 cycles (for patients with no measurable disease) or continues in the absence of disease progression or unacceptable toxicity (for patients with measurable disease).

RANDOMIZED PHASE II COMPONENT: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel IV over 1 hour once weekly and pazopanib hydrochloride PO QD for 2-3 weeks. Patients then receive concurrent paclitaxel IV over 1 hour once weekly and pazopanib hydrochloride PO QD for 6-7 weeks (or until radiation treatment is completed) and IMRT 5 days per week for 6.5 weeks (total of 66 Gy in 33 fractions). Beginning 25-31 days after the completion of IMRT, patients receive paclitaxel IV over 1 hour once weekly and pazopanib hydrochloride PO QD. Treatment repeats every 3 weeks for 4 cycles (for patients with no measurable disease) or continues in the absence of disease progression or unacceptable toxicity (for patients with measurable disease).

ARM II: Patients receive paclitaxel IV over 1 hour once weekly and placebo PO QD for 2-3 weeks. Patients then receive concurrent paclitaxel IV over 1 hour once weekly and placebo PO QD for 6-7 weeks (or until radiation treatment is completed) and IMRT 5 days per week for 6.5 weeks (total of 66 Gy in 33 fractions). Beginning 25-31 days after the completion of IMRT, patients receive paclitaxel IV over 1 hour once weekly and placebo PO QD. Treatment repeats every 3 weeks for 4 cycles (for patients with no measurable disease) or continues in the absence of disease progression or unacceptable toxicity (for patients with measurable disease).

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of anaplastic thyroid cancer (a diagnosis that is noted to be "consistent with anaplastic thyroid cancer" with the presence of a thyroid mass is acceptable)

  * Note: Tissue collection for central review is mandatory, but central review is not required for eligibility; due to the aggressiveness of this disease, treatment will be started prior to central review
* If there was a total or partial thyroidectomy completed within 3 months of enrollment, the surgical specimen must show the area of anaplastic thyroid cancer to be at least 1 cm in greatest dimension
* The following minimum diagnostic workup is required:

  * History/physical examination within 2 weeks prior to registration
  * Imaging of neck and brain (computed tomography [CT] scan or magnetic resonance imaging [MRI]) and chest/abdominal imaging (chest x-ray or chest CT scan, or full body positron emission tomography [PET]/CT are acceptable) within 4 weeks prior to registration
  * Note: The CT scan of the neck must be done with contrast or if an MRI is done, with gadolinium; therefore, the CT portion of a full body PET/CT has to be a high resolution CT to be acceptable for eligibility
  * Abdominal imaging must cover the liver and adrenal glands; therefore, separate imaging is not required if these areas are covered by a chest CT scan
  * Electrocardiogram within 10 days prior to registration
* Zubrod performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (within 10 days prior to registration on study)
* Platelets >= 100,000 cells/mm^3 (within 10 days prior to registration on study)
* Hemoglobin (Hgb) >= 9.0 g/dl (within 10 days prior to registration on study) (Note: the use of transfusion or other intervention to achieve Hgb >= 9.0 g/dL is acceptable)
* Total bilirubin < 1.5 x institutional upper limit of normal (ULN) (except for patients with Gilbert's syndrome and elevations of indirect bilirubin) (within 10 days prior to registration)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 x institutional ULN (within 10 days prior to registration); Note: patients who have both bilirubin > ULN and AST/ALT > ULN are not eligible (unless they have Gilbert's syndrome and elevations of indirect bilirubin)
* Spot urine protein to creatinine ratio (UPCR) < 1 or a 24-hour urine protein collection < 1 gm within 10 days prior to registration
* Creatinine < 1.5 mg/dL or within normal institutional limits within 10 days prior to registration; Note: if neither criteria is met, the creatinine clearance must be > 50 mL/min/1.73 m^2 per either the Cockcroft-Gault equation, Jeliffe method, or 12- or 24-hour urine collection
* Serum electrolytes including sodium, potassium, blood urea nitrogen (BUN), creatinine, glucose, magnesium, phosphate, and calcium within 10 days prior to registration
* Documentation of the patient's history of corrected QT interval (QTc) prolongation, family history of prolonged QTc, and relevant cardiac disease within 10 days prior to registration
* Evaluation of the patient's medications within 10 days prior to registration with attempt to change any medication that affects cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)
* Blood pressure =< 140/90 within 10 days of registration (must be taken and recorded by a health care professional); Note: if the systolic blood pressure is > 140 and/or diastolic blood pressure is > 90 at the time of registration, the patient's blood pressure must be controlled; systolic blood pressure must be < 140 and diastolic blood pressure must be < 90 on at least 2 separate measurements prior to the start of treatment, and the treating physician must believe that this is feasible in order to enroll the patient
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) within 1.2 x the upper limit of normal within 10 days prior to registration unless the patient is receiving coumadin and has a stable INR that is in range for the desired level of anticoagulation
* Negative pregnancy test (serum or urine) within 10 days of registration in women of child-bearing potential
* Women of childbearing potential and male participants who are sexually active must agree to practice adequate contraception during treatment and for 6 months post-treatment
* The patient must provide study specific informed consent prior to study entry

Exclusion Criteria:

* Known active invasive malignancy (except for non-melanomatous skin cancer or anaplastic thyroid cancer; the presence of prostate cancer confined to the prostate with a prostate-specific antigen [PSA] =< 1 ng/mL for more than 6 months also is allowed)
* Prior systemic chemotherapy for anaplastic thyroid cancer

  * Patients who have had chemotherapy or radiotherapy within 4 weeks of registration (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered > 4 weeks previously
  * Patients receiving other investigational agents
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Patients with any of the following cardiovascular conditions within the past 6 months:

  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * Admission for unstable angina
  * Myocardial Infarction
  * Cardiac angioplasty or stenting
  * Coronary artery bypass graft surgery
  * Pulmonary embolism, untreated deep venous thrombosis (DVT), or DVT which has been treated with therapeutic anticoagulation for less than 6 weeks
  * Arterial thrombosis
  * Symptomatic peripheral vascular disease
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; Note: a patient who has a history of class III heart failure and is asymptomatic on treatment may be considered eligible for the study
* Certain medications that are associated with a risk for QTc prolongation and/or torsades de pointes, although not prohibited, should be avoided or replaced with medications that do not carry these risks, if possible
* Patients who require heparin (other than low-molecular weight heparin)
* Patients with any condition that may impair the ability to absorb oral medications/investigational product including:

  * Prior surgical procedures affecting absorption including, but not limited to, major resection of stomach or small bowel
  * Active peptic ulcer disease
  * Malabsorption syndrome
* Patients with any condition that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, including:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesions
  * Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other gastrointestinal conditions which increase the risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
* History of hemoptysis within 30 days of registration; Note: patients who have minimal bleeding from the mouth, which is clearly not related to a source in the lungs, i.e., surgery such as a non-lung biopsy, are eligible only after good hemostasis has been documented
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Prior allergic reaction to the study drug(s) involved in this protocol
* QTc prolongation defined as a QTc interval >= 480 msecs or other significant electrocardiogram (EKG) abnormalities are ineligible; Note: if unsure about EKG abnormality, the treating physician should discuss this with Drs. Sherman or Bible
* Known brain metastasis
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with pazopanib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Certain medications that act through the cytochrome P450 (CYP450) system are specifically prohibited in patients receiving pazopanib and others should be avoided or administered with extreme caution

  * Strong inhibitors of CYP3A4 such as ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole may increase pazopanib concentrations and are prohibited; although, in exceptional circumstances, they may be administered in conjunction with lowering the dose of pazopanib by 50% of what would otherwise be administered; grapefruit juice is also an inhibitor of CYP450 and should not be taken with pazopanib
  * Strong inducers of CYP3A4, such as rifampin, may decrease pazopanib concentrations, are strictly prohibited
  * Medications that have narrow therapeutic windows and are substrates of CYP3A4, cytochrome P450, family 2, subfamily D, polypeptide 6 (CYP2D6), or cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8) should be avoided and, if necessary, administered with caution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-10-28 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Sherman, Principal Investigator — NRG Oncology
Locations (130):
- United States (130):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Billings Clinic Cancer Center, Billings, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Sherman EJ, Harris J, Bible KC, Xia P, Ghossein RA, Chung CH, Riaz N, Gunn GB, Foote RL, Yom SS, Wong SJ, Koyfman SA, Dzeda MF, Clump DA, Khan SA, Shah MH, Redmond K, Torres-Saavedra PA, Le QT, Lee NY. Radiotherapy and paclitaxel plus pazopanib or placebo in anaplastic thyroid cancer (NRG/RTOG 0912): a randomised, double-blind, placebo-controlled, multicentre, phase 2 trial. Lancet Oncol. 2023 Feb;24(2):175-186. doi: 10.1016/S1470-2045(22)00763-X. Epub 2023 Jan 18. PMID 36681089

RESULTS

PARTICIPANT FLOW:
Groups:
- (Run-in 1) Pazopanib, Paclitaxel, IMRT: Pre-Intensity-modulated radiation therapy (IMRT) pazopanib 800 mg oral daily and paclitaxel 80 mg/m^2 IV weekly for 2-3 weeks.
  Concurrent pazopanib 400 mg oral daily, paclitaxel 50 mg/m^2 IV weekly during 6.5 weeks of IMRT.
  Post-concurrent pazopanib 800 mg oral daily and paclitaxel 60 mg/m^2 IV weekly, starting 4 weeks after IMRT for 12 weeks if no evidence of disease or until progression or significant toxicity if evidence of disease.
- (Run-in 2) Pazopanib, Paclitaxil, IMRT: Pre-IMRT pazopanib 600 mg suspension oral daily and paclitaxel 80 mg/m^2 IV weekly for 2-3 weeks.
  Concurrent pazopanib 300 mg suspension oral daily, paclitaxel 50 mg/m^2 IV weekly during 6.5 weeks of IMRT.
- (Run-in 3) Pazopanib, Paclitaxel, IMRT; (Phase II) Pazopanib, Paclitaxel, IMRT: Pre-IMRT pazopanib 400 mg suspension oral daily and paclitaxel 80 mg/m^2 IV weekly for 2-3 weeks.
  Concurrent pazopanib 300 mg suspension oral daily, paclitaxel 50 mg/m^2 IV weekly during 6.5 weeks of IMRT.
- (Phase II) Placebo, Paclitaxel, IMRT: Pre-IMRT placebo 400 mg suspension oral daily and paclitaxel 80 mg/m^2 IV weekly for 2-3 weeks.
  Concurrent placebo 300 mg suspension oral daily, paclitaxel 50 mg/m^2 IV weekly during 6.5 weeks of IMRT.
Period: Overall Study
Arm/Group | (Run-in 1) Pazopanib, Paclitaxel, IMRT | (Run-in 2) Pazopanib, Paclitaxil, IMRT | (Run-in 3) Pazopanib, Paclitaxel, IMRT | (Phase II) Pazopanib, Paclitaxel, IMRT | (Phase II) Placebo, Paclitaxel, IMRT
Started | 11 | 11 | 12 | 42 | 47
Eligible | 11 | 10 | 11 | 36 | 35
Eligible and Started Study Treatment | 11 | 10 | 11 | 36 | 34
Eligible and Response Assessed | 0 | 0 | 0 | 23 | 27
Completed (Participants contributing data to results are considered to have completed the study) | 11 | 10 | 11 | 36 | 35
Not Completed | 0 | 1 | 1 | 6 | 12
Not completed — Protocol Violation | 0 | 1 | 1 | 6 | 12

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- (Run-in 1) Pazopanib, Paclitaxel, IMRT: Pre-IMRT pazopanib 800 mg oral daily and paclitaxel 80 mg/m^2 IV weekly for 2-3 weeks.
  Concurrent pazopanib 400 mg oral daily, paclitaxel 50 mg/m^2 IV weekly during 6.5 weeks of IMRT.
  Post-concurrent pazopanib 800 mg oral daily and paclitaxel 60 mg/m^2 IV weekly, starting 4 weeks after IMRT for 12 weeks if no evidence of disease or until progression or significant toxicity if evidence of disease.
  Intensity-Modulated Radiation Therapy: 33 fractions over 6.5 weeks, 5 fractions per week, 2 Gray per fraction to total dose of 66 Gy
- Total: Total of all reporting groups
Arm/Group | (Run-in 1) Pazopanib, Paclitaxel, IMRT | (Run-in 2) Pazopanib, Paclitaxil, IMRT | (Run-in 3) Pazopanib, Paclitaxel, IMRT | (Phase II) Pazopanib, Paclitaxel, IMRT | (Phase II) Placebo, Paclitaxel, IMRT | Total
Number analyzed (Participants) | 11 | 10 | 11 | 36 | 35 | 103
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 | 0 | 0 | 0 | 5 | 4 | 9
  50-59 | 3 | 1 | 1 | 5 | 7 | 17
  60-69 | 4 | 5 | 7 | 19 | 14 | 49
  ≥ 70 | 4 | 4 | 3 | 7 | 10 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 4 | 18 | 19 | 52
  Male | 7 | 3 | 7 | 18 | 16 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 1 | 3 | 7
  Not Hispanic or Latino | 8 | 10 | 10 | 29 | 24 | 81
  Unknown or Not Reported | 1 | 0 | 0 | 6 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 2 | 0 | 1 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 2 | 2 | 4
  White | 9 | 10 | 10 | 23 | 25 | 77
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 8 | 6 | 14
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 6 | 7 | 7 | 17 | 15 | 52
    1 | 4 | 3 | 4 | 17 | 16 | 44
    2 | 1 | 0 | 0 | 2 | 4 | 7
Prior surgery for study cancer [Count of Participants; unit: Participants] — Thyroidectomy is the surgical removal of all or part of the thyroid gland. Total thyroidectomy indicates that the entire thyroid gland was removed and partial thyroidectomy indicates that only part of the thyroid gland was removed.
  Participants
    None | 3 | 3 | 4 | 14 | 16 | 40
    Total thyroidectomy | 6 | 6 | 5 | 15 | 11 | 43
    Partial thyroidectomy | 2 | 1 | 2 | 7 | 8 | 20
T stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the size and/or extent of the main tumor. T4a = Intrathyroidal anaplastic carcinoma-surgically resectable. T4b = Extrathyroidal anaplastic carcinoma-surgically unresectable.
  Participants
    T4a | 4 | 2 | 1 | 11 | 12 | 30
    T4b | 7 | 8 | 10 | 25 | 23 | 73
N stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 7th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. N0 = No regional lymph node metastasis; N1a = Metastasis to Level VI (pretracheal, paratracheal, and prelaryngeal/Delphian lymph nodes); N1b = Metastasis to unilateral, bilateral, or contralateral cervical or superior mediastinal lymph nodes; NX = Lymph node status cannot be assessed.
  Participants
    N0 | 5 | 0 | 1 | 8 | 6 | 20
    N1a | 0 | 4 | 2 | 10 | 5 | 21
    N1b | 6 | 6 | 8 | 14 | 23 | 57
    NX | 0 | 0 | 0 | 4 | 1 | 5
M stage [Count of Participants; unit: Participants] — Distant metastasis stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the spread of the cancer to organs and tissues in other parts of the body. M0 = No distant metastasis; M1 = Distant metastasis; MX = Distant metastasis cannot be assessed.
  Participants
    M0 | 4 | 7 | 4 | 19 | 21 | 55
    M1 | 4 | 3 | 6 | 13 | 13 | 39
    Mx | 3 | 0 | 1 | 4 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: (Phase II) Overall Survival
Description: Overall survival time is defined as time from randomization to the date of death (failure) from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. One-year rates are provided. Analysis occurred after all eligible participants were potentially followed for 3 years.
Time Frame: From randomization to last follow-up.Maximum follow-up for phase II participants at time of analysis was 4.2 years.
Population: Eligible participants on phase II arms
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | (Phase II) Pazopanib, Paclitaxel, IMRT | (Phase II) Placebo, Paclitaxel, IMRT
Number analyzed (Participants) | 36 | 35
percentage of participants | 37.1 [21.1 to 53.2] | 29.0 [13.2 to 44.8]
Statistical Analysis 1: Comparison: (Phase II) Pazopanib, Paclitaxel, IMRT vs (Phase II) Placebo, Paclitaxel, IMRT; Assuming hazard ratio (pazopanib/placebo) of 0.625 (1-year 19% vs. 35.4%), 1-sided alpha 0.15, logrank test, 80% power, 1 interim analysis, required 71 deaths in 79 eligible patients (88 allowing 10% ineligible) in original design. The protocol was amended for phase II final analysis to be performed after all phase II eligible participants were potentially followed for 3 years with 1-sided alpha 0.1379, providing 77% power. See Limitations and Caveats; Test type: Superiority; p = 0.2831, Log Rank — One-sided significance level = 0.1379; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.52 to 1.43] — Reference arm = placebo

2. Primary Outcome: (Phase I) Number of Participants With Treatment-related Grade 4 Hemorrhage, Grade 4 Febrile Neutropenia, or Grade 5 Adverse Event (AE), or Discontinuation of Treatment Due to Toxicity [Adverse Events of Concern (AEC)]
Description: Common Terminology Criteria for AEs (version 4.0) grades AE severity from 1=mild to 5=death. Discontinuation of treatment due to toxicity is defined as < 75% of planned radiation therapy delivered. "Treatment-related" = definitely, probably, or possibly related to treatment. A single run-in arm was originally planned, but additional run-in arms were added due to amendments to the protocol regimen unrelated to toxicities. A two-stage design based on the binomial distribution was used in which the 1st stage analyzes the run-in arm and the 2nd stage analyzes run-in and phase II pazopanib arm participants combined. Because there were multiple run-in arms, only the last is used in the 2nd stage analysis. 1st stage: If ≤4 of 9 participants experience AEC, then conclude treatment is safe. 2nd stage: If ≤8 of 24 participants experience AEC, then conclude treatment safe. Otherwise conclude the treatment is too toxic. Summary data is provided here, see AE Module for specific AE data.
Time Frame: From registration to last follow-up. Maximum follow-up for run-in and phase II participants at time of analysis was 7.4 years.
Population: First nine eligible participants in run-in each arm and first 15 eligible participants in phase II pazopanib arm.
Measure: Count of Participants; unit: Participants
Groups:
- (Run-in 1) Pazopanib, Paclitaxel, IMRT: Pre-IMRT pazopanib 800 mg oral daily and paclitaxel 80 mg/m^2 IV weekly for 2-3 weeks.
  Concurrent pazopanib 400 mg oral daily, paclitaxel 50 mg/m^2 IV weekly during 6.5 weeks of IMRT.
  Post-concurrent pazopanib 800 mg oral daily and paclitaxel 60 mg/m^2 IV weekly, starting 4 weeks after IMRT for 12 weeks if no evidence of disease or until progression or significant toxicity if evidence of disease.
- (Phase II) Pazopanib, Paclitaxel, IMRT: Pre-IMRT pazopanib 400 mg suspension oral daily and paclitaxel 80 mg/m^2 IV weekly for 2-3 weeks.
  Concurrent pazopanib 300 mg suspension oral daily, paclitaxel 50 mg/m^2 IV weekly during 6.5 weeks of IMRT.
  Intensity-Modulated Radiation Therapy: 33 fractions over 6.5 weeks, 5 fractions per week, 2 Gray per fraction to total dose of 66 Gy
Arm/Group | (Run-in 1) Pazopanib, Paclitaxel, IMRT | (Run-in 2) Pazopanib, Paclitaxil, IMRT | (Run-in 3) Pazopanib, Paclitaxel, IMRT | (Phase II) Pazopanib, Paclitaxel, IMRT
Number analyzed (Participants) | 9 | 9 | 9 | 15
Participants | 0 | 0 | 2 | 0

3. Secondary Outcome: (Phase II) Local-regional Control
Description: Local-regional failure is defined as local-regional relapse/progression in the thyroid bed or regional lymph nodes. Time to local-regional failure is defined as time from randomization to the date of first local-regional recurrence, last known follow-up (censored), or death without local recurrence (competing risk). Failure rates are estimated using the cumulative incidence method. The protocol specifies 6- and 12-month estimates to be reported and for the full distributions of failure times to be compared between the arms. Analysis occurred after all eligible participants were potentially followed for 3 years.
Time Frame: From randomization to last follow-up.Maximum follow-up for phase II participants at time of analysis was 4.2 years. (Statistical analysis compares full distributions therefore all available follow-up was used.)
Population: Eligible participants on phase II arms
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | (Phase II) Pazopanib, Paclitaxel, IMRT | (Phase II) Placebo, Paclitaxel, IMRT
Number analyzed (Participants) | 36 | 35
percentage of participants
  6 months | 20.0 [8.6 to 34.8] | 27.3 [13.3 to 43.3]
  1 year | 28.6 [14.6 to 44.3] | 33.6 [17.9 to 50.0]
Statistical Analysis 1: Comparison: (Phase II) Pazopanib, Paclitaxel, IMRT vs (Phase II) Placebo, Paclitaxel, IMRT; Test type: Superiority; p = 0.6880, Log Rank; One-sided significance level = 0.15; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.55 to 2.67] — Reference arm = placebo

4. Secondary Outcome: (Phase II) Percentage of Participants With Treatment-related Grade 4 Hemorrhage, Grade 4 Febrile Neutropenia, or Grade 5 Adverse Event, or Discontinuation of Treatment Due to Toxicity [Adverse Events of Concern]
Description: Common Terminology Criteria for Adverse Events (CTCAE, v. 4.0) grades adverse event severity from 1=mild to 5=death. Discontinuation of treatment due to toxicity is defined as < 75% of planned radiation therapy delivered. Adverse events rated as definitely, probably, or possibly related to treatment were considered treatment-related. Summary data is provided in this outcome measure.; See Adverse Events Module for specific adverse event data.
Time Frame: From start of treatment to last follow-up.Maximum follow-up for phase II participants at time of analysis was 4.2 years.
Population: Eligible phase II participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | (Phase II) Pazopanib, Paclitaxel, IMRT | (Phase II) Placebo, Paclitaxel, IMRT
Number analyzed (Participants) | 36 | 34
percentage of participants | 2.8 [0.1 to 14.5] | 11.8 [3.3 to 27.5]
Statistical Analysis 1: Comparison: (Phase II) Pazopanib, Paclitaxel, IMRT vs (Phase II) Placebo, Paclitaxel, IMRT; Test type: Superiority; p = 0.1921, Fisher Exact — Two-sided significance level = 0.05

5. Secondary Outcome: (Phase II) Percentage of Participants With Treatment-related Grade 3 or 4 Adverse Events Other Than Grade 4 Hemorrhage or Grade 4 Febrile Neutropenia [Not Adverse Events of Concern]
Description: Common Terminology Criteria for Adverse Events (CTCAE, v. 4.0) grades adverse event severity from 1=mild to 5=death. Adverse events rated as definitely, probably, or possibly related to treatment were considered treatment-related. Summary data is provided in this outcome measure.; See Adverse Events Module for specific adverse event data.
Time Frame: From start of treatment to last follow-up.Maximum follow-up for phase II participants at time of analysis was 4.2 years.
Population: Eligible phase II participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | (Phase II) Pazopanib, Paclitaxel, IMRT | (Phase II) Placebo, Paclitaxel, IMRT
Number analyzed (Participants) | 36 | 34
percentage of participants | 86.1 [70.5 to 95.3] | 85.3 [68.9 to 95.0]
Statistical Analysis 1: Comparison: (Phase II) Pazopanib, Paclitaxel, IMRT vs (Phase II) Placebo, Paclitaxel, IMRT; Test type: Superiority; p = 1.00, Fisher Exact — Two-sided significance level = 0.05

6. Secondary Outcome: (Phase II) Percentage of Participants With Complete or Partial Response of the Primary Site After Chemoradiation Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Complete Response: Disappearance of all target lesions; Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 2-4 weeks after treatment (approximately week 10-14)
Population: Eligible participants on phase II arms that with response evaluated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | (Phase II) Pazopanib, Paclitaxel, IMRT | (Phase II) Placebo, Paclitaxel, IMRT
Number analyzed (Participants) | 23 | 27
percentage of participants | 30.4 [13.2 to 52.9] | 33.3 [16.5 to 54.0]
Statistical Analysis 1: Comparison: (Phase II) Pazopanib, Paclitaxel, IMRT vs (Phase II) Placebo, Paclitaxel, IMRT; Test type: Superiority; p = 1.00, Fisher Exact; Two-sided significance level = 0.05

ADVERSE EVENTS:
Time Frame: Weekly pre-IMRT and during IMRT, 2 weeks after IMRT, every months for years 1-2, every 6 months for year 3, then annually. Maximum follow-up time was 7.4 years for run-in arms and 4.2 years for phase II arms.
Arm/Group | (Run-in 1) Pazopanib, Paclitaxel, IMRT | (Run-in 2) Pazopanib, Paclitaxil, IMRT | (Run-in 3) Pazopanib, Paclitaxel, IMRT | (Phase II) Pazopanib, Paclitaxel, IMRT | (Phase II) Placebo, Paclitaxel, IMRT
All-Cause Mortality (participants affected / at risk) | 9/11 | 10/10 | 11/11 | 31/36 | 30/34
Serious Adverse Events (participants affected / at risk) | 9/11 | 6/10 | 8/11 | 28/36 | 22/34
Other Adverse Events (participants affected / at risk) | 10/11 | 10/10 | 11/11 | 36/36 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (Run-in 1) Pazopanib, Paclitaxel, IMRT (N=11) | (Run-in 2) Pazopanib, Paclitaxil, IMRT (N=10) | (Run-in 3) Pazopanib, Paclitaxel, IMRT (N=11) | (Phase II) Pazopanib, Paclitaxel, IMRT (N=36) | (Phase II) Placebo, Paclitaxel, IMRT (N=34)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 4 | 1 | 6 | 2
Esophageal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Death NOS (General disorders) | 1 | 0 | 0 | 0 | 0
Fever (General disorders) | 2 | 0 | 1 | 1 | 2
Neck edema (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Lung infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1 | 3 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2 | 0 | 0
Alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 1 | 1
Investigations - Other (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 2 | 3 | 3 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 4 | 2
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 4 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 3 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 2
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 4 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | (Run-in 1) Pazopanib, Paclitaxel, IMRT (N=11) | (Run-in 2) Pazopanib, Paclitaxil, IMRT (N=10) | (Run-in 3) Pazopanib, Paclitaxel, IMRT (N=11) | (Phase II) Pazopanib, Paclitaxel, IMRT (N=36) | (Phase II) Placebo, Paclitaxel, IMRT (N=34)
Anemia (Blood and lymphatic system disorders) | 8 | 6 | 6 | 15 | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 1 | 1 | 4
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Endocrine disorders - Other (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 4 | 1
Blurred vision (Eye disorders) | 1 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 3 | 3 | 8 | 10
Diarrhea (Gastrointestinal disorders) | 8 | 5 | 0 | 16 | 6
Dry mouth (Gastrointestinal disorders) | 5 | 8 | 5 | 17 | 15
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 4
Dysphagia (Gastrointestinal disorders) | 9 | 7 | 10 | 28 | 24
Esophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1
Esophageal stenosis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 | 0 | 1 | 8 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 6 | 7 | 7 | 18 | 16
Nausea (Gastrointestinal disorders) | 6 | 7 | 6 | 20 | 22
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1 | 4 | 5
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 3
Vomiting (Gastrointestinal disorders) | 5 | 4 | 3 | 10 | 13
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 2 | 0 | 4 | 2
Fatigue (General disorders) | 10 | 9 | 9 | 26 | 24
Fever (General disorders) | 5 | 0 | 3 | 3 | 5
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 0 | 8 | 2
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 2
Localized edema (General disorders) | 1 | 0 | 0 | 1 | 0
Neck edema (General disorders) | 1 | 1 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 1 | 1 | 0
Pain (General disorders) | 2 | 2 | 1 | 6 | 10
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 | 0 | 0 | 2 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 1 | 2
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Mucosal infection (Infections and infestations) | 1 | 1 | 0 | 2 | 3
Skin infection (Infections and infestations) | 1 | 2 | 1 | 2 | 2
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 7 | 10 | 8 | 22 | 26
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 6 | 8 | 5 | 17 | 3
Alkaline phosphatase increased (Investigations) | 5 | 4 | 1 | 10 | 2
Aspartate aminotransferase increased (Investigations) | 7 | 7 | 4 | 18 | 4
Blood bilirubin increased (Investigations) | 5 | 3 | 1 | 8 | 1
Creatinine increased (Investigations) | 1 | 0 | 2 | 2 | 4
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0 | 1 | 2
GGT increased (Investigations) | 1 | 0 | 0 | 1 | 1
INR increased (Investigations) | 2 | 1 | 0 | 0 | 2
Investigations - Other (Investigations) | 1 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 8 | 1 | 2 | 15 | 12
Neutrophil count decreased (Investigations) | 4 | 4 | 2 | 13 | 2
Platelet count decreased (Investigations) | 6 | 3 | 0 | 9 | 3
Weight loss (Investigations) | 6 | 5 | 4 | 10 | 12
White blood cell decreased (Investigations) | 8 | 6 | 4 | 17 | 6
Anorexia (Metabolism and nutrition disorders) | 2 | 5 | 3 | 11 | 12
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 3 | 5 | 6
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 5 | 3 | 11 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 6 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 6 | 3 | 10 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 6 | 3 | 12 | 9
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 7 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 4 | 3
Hyponatremia (Metabolism and nutrition disorders) | 5 | 3 | 2 | 12 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 2 | 1 | 4 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 0 | 2 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 3
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 14 | 10
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 7 | 1 | 1 | 4 | 2
Dysgeusia (Nervous system disorders) | 3 | 5 | 2 | 14 | 10
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 2 | 0 | 2 | 5
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Movements involuntary (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 4
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 4 | 2 | 8 | 4
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 2 | 9
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 2 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 1 | 6
Personality change (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 2 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 1 | 0 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 2 | 6 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1 | 7 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 12 | 13
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 5 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3 | 2 | 5
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2 | 3 | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 4 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 7 | 2 | 4 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 3 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 2 | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 10 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 2 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 9 | 4 | 6 | 13 | 16
Hypotension (Vascular disorders) | 1 | 0 | 0 | 7 | 3
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 4

LIMITATIONS AND CAVEATS:
One run-in arm was originally planned; more run-in arms added due to amendments to the protocol regimen unrelated to toxicities. In addition, due to higher than projected rates of ineligibility and consent withdrawals, phase II final analysis was amended to be time-driven (3 years of potential follow-up for all eligible phase II participants) instead of event driven (71 deaths of eligible phase II participants), reducing power from 80% (one-sided alpha 0.15) to 77% (one-sided alpha 0.1379),

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT01236547/Prot_SAP_000.pdf